CLINICAL TRIAL: NCT05022914
Title: Prostate-Specific Membrane Antigen (PSMA) Guided Approach for bIoCHEmical Relapse After Prostatectomy- A Prospective Observational Study-PSICHE
Brief Title: PSMA Guided Approach for bIoCHEmical Relapse After Prostatectomy-PSICHE
Acronym: PSICHE
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Lorenzo Livi, Full Professor, Azienda Ospedaliero-Universitaria Careggi
Other Study IDs: PSICHE
Record Dates: First submitted 2021-08-16; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Prostate Cancer; Biochemical Relapse Fo Malignant Neoplasm of Prostate; Prostate Adenocarcinoma; Prostate Cancer Recurrent
Keywords: PSMA; 68Ga-PSMA PET/CT; PET/CT; Biochemical Relapse; micro-RNA; SBRT; Radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Panel of miRNA (miR-186, miR-26a, miR-374a, miR-410, miR-660)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Patients affected by biochemical relapse after radical prostatectomy undergoing staging PSMA-PET/CT and baseline blood sample for miRNA panel assessment.

SUMMARY:
This observational study was designed to evaluate progression free survival after PSMA-PET/CT based salvage approach for patients affected by biochemical relapse after radical prostatectomy.

DETAILED DESCRIPTION:
This is a prospective observational multicenter study including patients treated with upfront radical prostatectomy +/- postoperative prostate bed radiotherapy, with histological result of Prostate adenocarcinoma, affected by biochemical relapse (defined as PSA>/= 0.2 ng/ml) with a PSA at recurrence </=1 ng/ml. Patients will be staged with centralized 68 Ga- PSMA PET/CT and treated with a pre-defined approach based on 68 Ga-PSMA PET/CT findings.

The predefined approach will consist in the following flowchart:

1. In negative 68Ga-PSMA PET/CT or positive findings within prostate bed: Prostate bed RT
2. In 68Ga-PSMA PET/CT detecting pelvic nodal recurrence amenable with stereotactic body radiation therapy (SBRT) on all sites of disease: SBRT to all positive nodal disease.
3. In abdominal nodal or bone oligometastatic disease amenable with stereotactic body radiation therapy (SBRT) on all sites of disease: SBRT on all sites of disease
4. In abdominal nodal or bone metastatic disease (>3 lesions or non-amenable with SBRT) and/or visceral disease: ADT+/-other systemic therapies available for metastatic hormone sensitive pCa at physician discretion.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age >18
* Patient suitable for 68Ga-PSMA PET/CT re-staging according to clinical practice (Previous radical prostatectomy with histological result of Prostate adenocarcinoma +/- postoperative prostate bed radiotherapy (adjuvant or salvage setting), with a biochemical relapse defined as a PSA > 0.2 and <1

Exclusion Criteria:

* ADT administration within 6 months from study enrollment
* Persistent elevation of PSA after RP measured within 16 weeks from surgery (> 0.1 ng/ml)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer male patient
Study Population: Patient affected by biochemical recurrence after radical prostatectomy.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2024-01-19 (Estimated); Study Completion 2027-01-19 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 2 year
  PFS is defined as time from end of salvage treatment performed at first relapse to documented biochemical progression or radiological progression (or both), death from any cause or censoring at date of last follow-up.

SECONDARY OUTCOMES:
Overall Survival | 2 years
  Time between end of tailored treatment after 68Ga-PSMA PET/CT and death.
Cause-specific survival | 2 years
  Time between end of tailored treatment and death for prostate Cancer.
Radiological Progression Free Survival | 2 years
  The occurrence of any new lesion detectable with PSMA. PET/CT and/or any other molecular/radiological exam, which will be performed in case of biochemical or clinical progression.
Quality of Life | 2 years
  Record rate of patients with impaired quality of life measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-C30
Quality of Life | 2 years
  Record rate of patients with impaired quality of life measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-PR25
Management Change | 2 years
  Assess the proportion of management changes induced by positive PSMA PET/CT results.
Association between PSMA PET/CT Detection Rate and specific miRNA panel | 2 year
  Association between PSMA PET/CT Detection Rate and specific miRNA panel

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Livi, Prof., Principal Investigator — Azienda Ospedaliero-Universitaria Careggi
Locations (1):
- AOU Careggi Radiation Oncology Unit, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mottet N, Bellmunt J, Bolla M, Briers E, Cumberbatch MG, De Santis M, Fossati N, Gross T, Henry AM, Joniau S, Lam TB, Mason MD, Matveev VB, Moldovan PC, van den Bergh RCN, Van den Broeck T, van der Poel HG, van der Kwast TH, Rouviere O, Schoots IG, Wiegel T, Cornford P. EAU-ESTRO-SIOG Guidelines on Prostate Cancer. Part 1: Screening, Diagnosis, and Local Treatment with Curative Intent. Eur Urol. 2017 Apr;71(4):618-629. doi: 10.1016/j.eururo.2016.08.003. Epub 2016 Aug 25. PMID 27568654
- [Result] Thompson IM, Valicenti RK, Albertsen P, Davis BJ, Goldenberg SL, Hahn C, Klein E, Michalski J, Roach M, Sartor O, Wolf JS Jr, Faraday MM. Adjuvant and salvage radiotherapy after prostatectomy: AUA/ASTRO Guideline. J Urol. 2013 Aug;190(2):441-9. doi: 10.1016/j.juro.2013.05.032. Epub 2013 May 21. PMID 23707439
- [Result] Pisansky TM, Thompson IM, Valicenti RK, D'Amico AV, Selvarajah S. Adjuvant and Salvage Radiotherapy after Prostatectomy: ASTRO/AUA Guideline Amendment 2018-2019. J Urol. 2019 Sep;202(3):533-538. doi: 10.1097/JU.0000000000000295. Epub 2019 Aug 8. PMID 31042111
- [Result] Tendulkar RD, Agrawal S, Gao T, Efstathiou JA, Pisansky TM, Michalski JM, Koontz BF, Hamstra DA, Feng FY, Liauw SL, Abramowitz MC, Pollack A, Anscher MS, Moghanaki D, Den RB, Stephans KL, Zietman AL, Lee WR, Kattan MW, Stephenson AJ. Contemporary Update of a Multi-Institutional Predictive Nomogram for Salvage Radiotherapy After Radical Prostatectomy. J Clin Oncol. 2016 Oct 20;34(30):3648-3654. doi: 10.1200/JCO.2016.67.9647. PMID 27528718
- [Result] Cornford P, Bellmunt J, Bolla M, Briers E, De Santis M, Gross T, Henry AM, Joniau S, Lam TB, Mason MD, van der Poel HG, van der Kwast TH, Rouviere O, Wiegel T, Mottet N. EAU-ESTRO-SIOG Guidelines on Prostate Cancer. Part II: Treatment of Relapsing, Metastatic, and Castration-Resistant Prostate Cancer. Eur Urol. 2017 Apr;71(4):630-642. doi: 10.1016/j.eururo.2016.08.002. Epub 2016 Aug 31. PMID 27591931
- [Result] Afshar-Oromieh A, Holland-Letz T, Giesel FL, Kratochwil C, Mier W, Haufe S, Debus N, Eder M, Eisenhut M, Schafer M, Neels O, Hohenfellner M, Kopka K, Kauczor HU, Debus J, Haberkorn U. Diagnostic performance of 68Ga-PSMA-11 (HBED-CC) PET/CT in patients with recurrent prostate cancer: evaluation in 1007 patients. Eur J Nucl Med Mol Imaging. 2017 Aug;44(8):1258-1268. doi: 10.1007/s00259-017-3711-7. Epub 2017 May 12. PMID 28497198
- [Result] Calais J, Ceci F, Eiber M, Hope TA, Hofman MS, Rischpler C, Bach-Gansmo T, Nanni C, Savir-Baruch B, Elashoff D, Grogan T, Dahlbom M, Slavik R, Gartmann J, Nguyen K, Lok V, Jadvar H, Kishan AU, Rettig MB, Reiter RE, Fendler WP, Czernin J. 18F-fluciclovine PET-CT and 68Ga-PSMA-11 PET-CT in patients with early biochemical recurrence after prostatectomy: a prospective, single-centre, single-arm, comparative imaging trial. Lancet Oncol. 2019 Sep;20(9):1286-1294. doi: 10.1016/S1470-2045(19)30415-2. Epub 2019 Jul 30. PMID 31375469
- [Result] Ost P, Bossi A, Decaestecker K, De Meerleer G, Giannarini G, Karnes RJ, Roach M 3rd, Briganti A. Metastasis-directed therapy of regional and distant recurrences after curative treatment of prostate cancer: a systematic review of the literature. Eur Urol. 2015 May;67(5):852-63. doi: 10.1016/j.eururo.2014.09.004. Epub 2014 Sep 17. PMID 25240974
- [Result] Deandreis D, Guarneri A, Ceci F, Lillaz B, Bartoncini S, Oderda M, Nicolotti DG, Pilati E, Passera R, Zitella A, Bello M, Parise R, Carlevato R, Ricardi U, Gontero P. 68Ga-PSMA-11 PET/CT in recurrent hormone-sensitive prostate cancer (HSPC): a prospective single-centre study in patients eligible for salvage therapy. Eur J Nucl Med Mol Imaging. 2020 Nov;47(12):2804-2815. doi: 10.1007/s00259-020-04809-8. Epub 2020 Apr 20. PMID 32314028
- [Result] Erdmann K, Kaulke K, Thomae C, Huebner D, Sergon M, Froehner M, Wirth MP, Fuessel S. Elevated expression of prostate cancer-associated genes is linked to down-regulation of microRNAs. BMC Cancer. 2014 Feb 11;14:82. doi: 10.1186/1471-2407-14-82. PMID 24517338
- [Result] D'Angelillo RM, Francolini G, Ingrosso G, Ravo V, Triggiani L, Magli A, Mazzeo E, Arcangeli S, Alongi F, Jereczek-Fossa BA, Pergolizzi S, Pappagallo GL, Magrini SM. Consensus statements on ablative radiotherapy for oligometastatic prostate cancer: A position paper of Italian Association of Radiotherapy and Clinical Oncology (AIRO). Crit Rev Oncol Hematol. 2019 Jun;138:24-28. doi: 10.1016/j.critrevonc.2019.03.014. Epub 2019 Apr 1. PMID 31092381
- [Result] Carrie C, Magne N, Burban-Provost P, Sargos P, Latorzeff I, Lagrange JL, Supiot S, Belkacemi Y, Peiffert D, Allouache N, Dubray BM, Servagi-Vernat S, Suchaud JP, Crehange G, Guerif S, Brihoum M, Barbier N, Graff-Cailleaud P, Ruffion A, Dussart S, Ferlay C, Chabaud S. Short-term androgen deprivation therapy combined with radiotherapy as salvage treatment after radical prostatectomy for prostate cancer (GETUG-AFU 16): a 112-month follow-up of a phase 3, randomised trial. Lancet Oncol. 2019 Dec;20(12):1740-1749. doi: 10.1016/S1470-2045(19)30486-3. Epub 2019 Oct 16. PMID 31629656
- [Derived] Francolini G, Banini M, Di Cataldo V, Detti B, Caini S, Loi M, Simontacchi G, Desideri I, Greto D, Valzano M, Roghi M, Serni S, Vaggelli L, Salvestrini V, Visani L, Becherini C, Olmetto E, Franzese C, Baldaccini D, Scorsetti M, Sollini M, Chiti A, Meattini I, Valicenti RK, Livi L. PSMA guided approach for bIoCHEmical relapse after prostatectomy- (PSICHE) trial (NCT05022914). Detection rate and treatment decision after 68Ga-PSMA PET/CT within a prospective study. Prostate. 2023 Sep;83(12):1201-1206. doi: 10.1002/pros.24579. Epub 2023 Jun 8. PMID 37290915
- [Derived] Francolini G, Di Cataldo V, Detti B, Simontacchi G, Loi M, Valzano M, Desideri I, Meattini I, Mangoni M, Livi L. Killing two birds with a stone: how to maximise benefit from metastasis-directed therapy and modern systemic treatment in oligometastatic hormone sensitive prostate cancer. Clin Exp Metastasis. 2022 Dec;39(6):841-843. doi: 10.1007/s10585-022-10187-2. Epub 2022 Oct 15. PMID 36242700